CLINICAL TRIAL: NCT03681353
Title: Impact of Reduced Cannabis Use on Functional Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00100100
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Cannabis; Cannabis Use
MeSH Terms: conditions — Marijuana Abuse | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Use Condition (Experimental): This arm includes six weeks of mobile contingency management treatment administered via a smart-phone based application (mobile CM), in which participants are provided monetary reinforcement for reducing cannabis use.
  Interventions: Behavioral: Mobile Contingency Management, active

INTERVENTIONS:
Behavioral: Mobile Contingency Management, active — Participants are provided monetary reinforcement for providing oral fluid test results that suggest they have reduced cannabis use.

SUMMARY:
Nearly 20 million Americans report use of cannabis in the past month, and heavy cannabis use has increased by nearly 60% in the U.S. since 2007. Heavy cannabis use is associated with lower educational attainment, reduced physical activity, and increased rates of addiction, unemployment, and neuropsychological deficits. Studies by the lab and others suggest that cannabis use is also associated with increased mental health symptoms and suicidal and nonsuicidal self-injury. In addition, cannabis is the illicit drug most strongly associated with drugged driving and traffic accidents, including fatal accidents. There is evidence that sustained abstinence from cannabis can lead to improvements in the functional outcomes of former users. However, he degree to which reductions in cannabis use might be associated with positive changes in functional outcomes is currently unknown. The overall objective of the present research is to use ecological momentary assessment (EMA), a real-time, naturalistic data collection method, to study the impact of reduced cannabis use on functional outcomes in heavy cannabis users. Contingency management (CM) will be used to promote reductions in frequency and quantity of cannabis use. CM is an intensive behavioral therapy that is highly effective at producing short-term reductions in illicit drug use. The investigators novel approach includes mobile technology to make CM more portable and feasible. The present research will use this technology in conjunction with state-of-the-art EMA methods to study the impact of reduced cannabis use on key functional outcomes. The investigators central hypothesis is that reductions in frequency and quantity of cannabis use will lead to positive changes in cannabis users' mental health, physical activity, working memory, health-related quality of life, and driving behavior.

DETAILED DESCRIPTION:
Nearly 20 million Americans report use of cannabis in the past month, and heavy cannabis use has increased by nearly 60% in the U.S. since 2007. Heavy cannabis use is associated with lower educational attainment, reduced physical activity, and increased rates of addiction, unemployment, and neuropsychological deficits. Studies by the lab and others suggest that cannabis use is also associated with increased mental health symptoms and suicidal and nonsuicidal self-injury. In addition, cannabis is the illicit drug most strongly associated with drugged driving and traffic accidents, including fatal accidents. While there is evidence that sustained abstinence can lead to improvements in the functional outcomes of former users, the degree to which reductions in cannabis use alone (i.e., in the absence of sustained abstinence) might be associated with positive changes in functional outcomes is currently unknown. This is a critical gap in the literature, as many clinical interventions for cannabis and other drugs are associated with decreases in frequency and quantity of use, but fail to achieve an effect on overall abstinence rates. The overall objective of the present research is to use ecological momentary assessment (EMA), a real-time, naturalistic data collection method, to prospectively study the impact of reduced cannabis use on functional outcomes in heavy cannabis users. EMA addresses several limitations of traditional assessment techniques by enhancing ecological validity, minimizing memory bias, and enabling examination of the impact of context on participants' behavior. Contingency management (CM) will be used to promote reductions in frequency and quantity of cannabis use. CM is an intensive behavioral therapy that is highly effective at producing short-term reductions in illicit drug use. Moreover, the investigators have recently developed a novel approach that leverages mobile technology and recent developments in cannabis testing to make CM for cannabis more portable and feasible. The investigators have pilot-tested this approach with heavy cannabis users and found that it is an acceptable and feasible method to reduce their cannabis use. The present research will use this technology in conjunction with state-of-the-art EMA methods to study the impact of reduced cannabis use on key functional outcomes. The investigators central hypothesis is that reductions in frequency and quantity of cannabis use will lead to positive changes in cannabis users' mental health, physical activity, working memory, health-related quality of life, and driving behavior. The rationale for this research is that it will provide the first and only real-time data concerning the potential impact of reductions in cannabis use on functional outcomes. As such, the findings from the present research will directly inform ongoing efforts to include reductions in illicit drug use as a valid, clinically-meaningful outcome measure in clinical trials of pharmacotherapies for the treatment of substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* cannabis use on ≥40 of past 90 days
* ability to speak and write fluent English
* 18-70 years of age
* willingness to attempt to temporarily reduce cannabis use

Exclusion Criteria:

* expect to have an unstable medication regimen during the study
* are currently receiving non-study CUD treatment
* meet criteria for serious mental illness (e.g., bipolar disorder, schizophrenia)
* become imprisoned
* become hospitalized for psychiatric reasons
* become pregnant
* report imminent risk for suicide or homicide
* meet criteria for a substance use disorder other than CUD or tobacco

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reduced Use Condition
Started | 25
Completed | 18
Not Completed | 7
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — withdrawn by PI | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Reduced Use Condition
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.95 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 5
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete the Baseline Assessment
Description: Adherence is defined as completing the baseline assessment
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Use Condition
Number analyzed (Participants) | 18
Participants | 18

2. Primary Outcome: Number of Participants Who Complete the 8-week Follow-up Assessment
Description: Adherence is defined as completing the 8-week follow-up assessment
Time Frame: 8- week follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Use Condition
Number analyzed (Participants) | 18
Participants | 18

3. Primary Outcome: Number of Participants Who Complete 1 or More Ecological Momentary Assessments (EMA) Per Day (Total ≥56) for the Duration of the 8-week EMA Protocol
Description: Adherence is defined as completing 1 or more EMA assessments per day (total ≥56) for the duration of the 8-week EMA protocol
Time Frame: 8 week follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Use Condition
Number analyzed (Participants) | 18
Participants | 8

4. Primary Outcome: Number of Participants Who Score Above Threshold on Treatment Acceptability Measure
Description: Acceptability of treatment will be measured by a questionnaire designed for use in this study. A single item measured acceptability of treatment, with a Likert scale (1-10) response in which 1=extremely unacceptable and 10=extremely acceptable. Threshold for acceptability is a score of 6 or greater.
Time Frame: 8-week posttreatment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Use Condition
Number analyzed (Participants) | 18
Participants | 18

5. Secondary Outcome: Number of Participants Who Have ≥ 50% Reduction in Frequency of Cannabis Use
Description: To evaluate if this milestone has been met, the investigators will calculate the percentage reduction in bioverified abstinent days by comparing the ad lib monitoring period to the mobile CM period.
Time Frame: Ad lib monitoring period (up to 2 weeks), 8-week posttreatment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Use Condition
Number analyzed (Participants) | 18
Participants | 12

6. Secondary Outcome: Average Number of Days Since Last Cannabis Use
Description: Investigators will use count-adjusted (i.e., negative binomial or Poisson) MLM to model the equivalent number of joints/gram smoked on a given day as a function of days since last use.
Time Frame: 8-week posttreatment visit
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Reduced Use Condition
Number analyzed (Participants) | 18
days | 6.95 (9.55)

7. Secondary Outcome: Number of Participants Who Have ≥ 50% Reduction in Quantity of Cannabis Use
Description: To evaluate if this milestone has been met, the investigators will calculate the percentage reduction in overall cannabis quantity by comparing the ad lib monitoring period to the mobile CM period.
Time Frame: Ad lib monitoring period (up to 2 weeks), 8-week posttreatment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Use Condition
Number analyzed (Participants) | 18
Participants | 18

ADVERSE EVENTS:
Time Frame: Adverse events were collected for approximately eight weeks, from informed consent signature to the post-treatment visit.
Arm/Group | Reduced Use Condition
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Use Condition (N=18)
Psychiatric inpatient hospitalization (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Use Condition (N=18)
Distress related to death in family (Psychiatric disorders) | 1 (1)
Broken arm (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03681353/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03681353/ICF_001.pdf